CLINICAL TRIAL: NCT05866497
Title: Relationship Between Periodontal Status and Cardio Ankle Vascular Index in Short-term Type 2 Diabetic or Systemically Healthy Patients With or Without Severe Periodontitis
Brief Title: Arterial Stiffness in Type 2 Diabetic Patients With Severe Periodontitis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gizem Torumtay Cin, assistant professor, Pamukkale University
Other Study IDs: 07.06.2022/09
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Coronary Heart Disease; Diabetes Mellitus, Type 2; Periodontitis; Arterial Stiffness
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- diabetes and periodontitis group (group 1): 35 subjects with type 2 diabetes and severe periodontitis were recruited in group 1.
  The clinical periodontal parameters taken are as follows:
  plaque index (PI), gingival index (GI), bleeding on brobing (BOP), probing depth (PD) and clinical attachment level (CAL).
  The present number of teeth in participants was recorded. Cardio-ankle vascular index (CAVI) was measured
  Interventions: Diagnostic Test: clinical periodontal measurements; Diagnostic Test: CAVI measurements
- diabetes and periodontally healthy (group 2): 34 subjects with type 2 diabetes and periodontally healthy were recruited in group 2.
  The clinical periodontal parameters taken are as follows:
  plaque index (PI), gingival index (GI), bleeding on brobing (BOP), probing depth (PD) and clinical attachment level (CAL).
  The present number of teeth in participants was recorded. Cardio-ankle vascular index (CAVI) was measured
  Interventions: Diagnostic Test: clinical periodontal measurements; Diagnostic Test: CAVI measurements
- systemically healthy and periodontitis (group 3): 32 systemically healthy subjects with severe periodontitis were recruited in group 3.
  The clinical periodontal parameters taken are as follows:
  plaque index (PI), gingival index (GI), bleeding on brobing (BOP), probing depth (PD) and clinical attachment level (CAL).
  The present number of teeth in participants was recorded. Cardio-ankle vascular index (CAVI) was measured
  Interventions: Diagnostic Test: clinical periodontal measurements; Diagnostic Test: CAVI measurements
- systemically healthy and periodontally healthy (group 4): 35 systemically and periodontally healthy subjects were recruited in group 4.
  The clinical periodontal parameters taken are as follows:
  plaque index (PI), gingival index (GI), bleeding on brobing (BOP), probing depth (PD) and clinical attachment level (CAL).
  The present number of teeth in participants was recorded. Cardio-ankle vascular index (CAVI) was measured
  Interventions: Diagnostic Test: clinical periodontal measurements; Diagnostic Test: CAVI measurements

INTERVENTIONS:
Diagnostic Test: clinical periodontal measurements — Periodontal parameters such as PI, GI, BOP, PD, and CAL were measured using the Williams periodontal probe (Hu-Friedy, Chicago IL). PD and CAL were calculated at six surfaces per tooth, whereas PI and GI were measured at four surfaces per tooth.
  The periodontal status of patients was determined based on the Classification of Periodontal and Peri-Implant Diseases and Conditions stated in 2017 World Workshop
Diagnostic Test: CAVI measurements — Arterial stiffness of the participants included in this study were assessed by CAVI index using VaSera (VS-1500N) CAVI device (Fukuda Denshi Co. Ltd., Tokyo, Japan) between both arms and ankles in a supine position.
  Right and left CAVI values were calculated separately.

SUMMARY:
Studies were found that a significant relationship between the severe periodontitis and increased CAVI values. While the exact mechanisms linking periodontitis, type 2 diabetes, and cardiovascular disease are not yet fully understood, it is clear that these diseases are interconnected. There are limited data in the literature evaluating the risk of atherosclerosis in diabetic individuals with periodontal disease. In our survey, we hypothesised that severe periodontitis may be a risk factor for the development of subclinical atherosclerosis among people with type 2 diabetes. Thus, we aimed to investigate the potential risk of subclinical atherosclerosis by using a new surrogate marker CAVI in severe periodontitis patients with short-term diabetes.

DETAILED DESCRIPTION:
Short-term diabetic subjects were selected from patients diagnosed with type 2 diabetes for less than 5 years recruited from those patients attending to the outpatient clinic at the Department of Endocrinology in University Hospital. Medical conditions of SH subjects were determined with detailed systemic examinations and biochemical analyses were performed in the Department of Endocrinology.

The periodontal status of patients was determined based on the Classification of Periodontal and Peri-Implant Diseases and Conditions stated in 2017 World Workshop. Periodontally health was considered if the volunteers have clinically healthy gingiva on an intact periodontium who had BOP < 10% and PD ≤ 3 mm, no sites with attachment loss, no radiographic sign of alveolar bone destruction and no history of periodontitis. Patients with severe periodontitis were defined if they had interdental CAL ≥ 5 mm, PD ≥ 6 mm and radiographic bone loss extending to the mid-third of the root or beyond.

Assessment of participants included in this study in terms of arterial stiffness was determined by CAVI index. Right and left CAVI values were calculated separately, and their mean value was used for the analysis. Besides the mean CAVI values, the CAVI values were categorized. CAVI ≥ 8 was considered conditionally pathological, while CAVI ≥ 9 was defined as pathologic.

Various metabolic variables of the participants were collected at baseline to eliminate previously reported confounding factors as being associated with periodontitis and arterial stiffness. The body mass index (BMI) was calculated by taking the weight, in kilograms divided by the height in meters squared. BMI ≥ 25 kg/m2 was defined as overweight and BMI ≥ 30 kg/m2 as obese. Waist circumference (WC) was also recorded. Medical conditions were analysed by hematologic results. Glycated haemoglobin (HbA1c) and fasting plasma glucose (FPG) were assessed for the glycemic control levels of the participants. Also, dyslipidaemia and hyperlipidaemia were evaluated by the measurements of low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglyceride (TRG) and total cholesterol (TK) levels. Systolic (SBP) and diastolic blood pressure (DBP) was measured and SBP ≥ 140 mmHg or DBP ≥ 90 mmHg was defined as hypertension and excluded from the study population. C-reactive protein (CRP) levels of the participants were also evaluated at the beginning of the study.

The power analyse of the study was performed for sample size calculation. Sample size was calculated using the G*Power software program (G*Power; Universitat, Dusseldorf, Germany) for α = 0.05 and f = 0.3. The analyses revealed that 32 subjects per group achieved a power of 80 % with 95% confidence.

The data were analysed with the SPSS 21 program (SPSS Inc., Chicago, IL). Continuous variables were presented as mean ± standard deviation and categorical variables as numbers and percentages. Shapiro-Wilk test was used to detect data's normality. For the comparison of the parameters of the study groups, One-way ANOVA test was used for normally distributed data while Kruskal-Wallis test was performed as non-parametric test. Chi-square test was used for the comparison of the categorical variables. Statistical significance value was considered as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* short-term type 2 diabetes mellitus diagnosis (<5 years) or systemically healthy subjects
* patients with severe periodontitis or periodontally healthy subjects

Exclusion Criteria:

* had vascular diabetic complications
* hypertensive and dyslipidaemic/hyperlipidaemic patients
* Smokers and ex-smokers
* pregnancy and lactation
* using systemic antibiotic or anti-inflammatory drugs in the 6 months before the start of the study
* history of past periodontal treatment within 6 months period
* ankle-branchial index (ABI) values less than 0.9
* obesity with BMI ≥ 30 kg/m2

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic subjects were selected from patients diagnosed with type 2 diabetes for less than 5 years recruited from those patients attending to the outpatient clinic at the Department of Endocrinology at Pamukkale University Hospital.
  Systemically healthy subjects were recruited from the patients who referred to Faculty of Dentistry in Pamukkale University for dental treatments. Medical conditions of systemically healthy subjects were determined with detailed systemic examinations and biochemical analyses were performed in the Department of Endocrinology at Pamukkale University Hospital.
  Patients with severe periodontitis or periodontally healthy subjects were selected from the patients who referred to the Periodontology Clinic in Faculty of Dentistry at Pamukkale University for periodontal examinations.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
CAVI measurements | at baseline
  mean CAVI values (m/s) in each study groups

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Torumtay Cin, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University Faculty of Dentistry, Denizli, Turkey (Türkiye)